CLINICAL TRIAL: NCT01721343
Title: MC1193: Collaborative Care to Preserve Performance in Cancer (COPE)
Brief Title: Collaborative Targeted Case Management in Improving Functional Status in Patients with Stage III-IV Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC1193; R01CA163803 (NIH); NCI-2012-01603 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-10-08; First posted 2012-11-05 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cognitive/functional Effects; Malignant Neoplasm; Pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Case Management; Physical Therapy Modalities; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (enhanced usual care) (Experimental): Patients undergo enhanced usual care comprising telephonic monitoring with monthly status reports provided to their oncology care teams for 6 months.
  Interventions: Behavioral: telephone-based intervention; Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: management of therapy complications; Procedure: assessment of therapy complications
- Arm II (enhanced usual care, RCM) (Experimental): Patients undergo enhanced usual care as in Arm I and participate in an individualized conditioning program delivered telephonically by the Fitness Care Manager (FCM) and adapted, as required, by a local physical therapist for 6 months.
  Interventions: Behavioral: telephone-based intervention; Other: case management; Procedure: physical therapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Other: educational intervention; Procedure: management of therapy complications; Procedure: assessment of therapy complications
- Arm III (enhanced usual, RCM, PCM) (Experimental): Patients undergo enhanced usual care as in Arm I, participate in an individualized conditioning program coordinated by the FCM as in Arm II, and receive optimized pain management through a nurse Pain Care Manager (PCM) for 6 months.
  Interventions: Behavioral: telephone-based intervention; Other: case management; Procedure: management of therapy complications; Procedure: physical therapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Other: educational intervention; Procedure: assessment of therapy complications

INTERVENTIONS:
Behavioral: telephone-based intervention — Undergo telephonic monitoring
Other: case management — Participate in an individualized conditioning program with an RCM
  Arms: Arm II (enhanced usual care, RCM); Arm III (enhanced usual, RCM, PCM)
Procedure: management of therapy complications — Undergo enhanced usual care with an RCM and PCM
  Other Names: complications of therapy, management of
  Arms: Arm III (enhanced usual, RCM, PCM)
Procedure: physical therapy — Participate in an individualized conditioning program with an RCM
  Other Names: physiotherapy
  Arms: Arm II (enhanced usual care, RCM); Arm III (enhanced usual, RCM, PCM)
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: management of therapy complications — Undergo enhanced usual care
  Other Names: complications of therapy, management of
  Arms: Arm I (enhanced usual care)
Procedure: assessment of therapy complications — Undergo enhanced usual care
  Arms: Arm I (enhanced usual care)
Other: educational intervention — Participate in an individualized conditioning program with an RCM
  Other Names: intervention, educational
  Arms: Arm II (enhanced usual care, RCM); Arm III (enhanced usual, RCM, PCM)
Procedure: management of therapy complications — Undergo enhanced usual care with an RCM
  Other Names: complications of therapy, management of
  Arms: Arm II (enhanced usual care, RCM)
Procedure: assessment of therapy complications — Undergo enhanced usual care with an RCM
  Arms: Arm II (enhanced usual care, RCM)
Procedure: assessment of therapy complications — Undergo enhanced usual care with an RCM and PCM
  Arms: Arm III (enhanced usual, RCM, PCM)

SUMMARY:
This randomized clinical trial studies collaborative targeted case management in improving functional status in patients with stage III-IV cancer. Collaborative targeted case management may improve functional mobility, improve quality of life, and reduce pain and health care utilization in patients with advanced cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the comparative effectiveness of the Collaborative Care to Preserve Performance in Cancer (COPE) trial arms in preserving functional mobility.

II. To assess the comparative cost-effectiveness and cost-utility of the COPE interventions.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients undergo enhanced usual care comprising telephonic monitoring with monthly status reports provided to their oncology care teams for 6 months.

ARM II: Patients undergo enhanced usual care as in Arm I and participate in an individualized conditioning program delivered telephonically by the Fitness Care Manager (FCM) and adapted, as required, by a local physical therapist for 6 months.

ARM III: Patients undergo enhanced usual care as in Arm I, participate in an individualized conditioning program coordinated by the FCM as in Arm II, and receive optimized pain management through a nurse Pain Care Manager (PCM) for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III or stage IV cancer
* Life expectancy > 6 months
* Ambulatory Post Acute Care (APC) score between 53 and 66
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Have working phone to communicate with study team
* Fluent in English
* Sufficient auditory acuity
* Intact cognitive status

Exclusion Criteria:

* Patient is within 2 months of a major surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
Functional mobility, as measured by the change in the Activity Measure for Post Acute Care (AM PAC) Computer Adaptive Test (CAT) from baseline [6 months] | From baseline to 6 months
  The mean change in the Ambulatory Post-Acute Care Basic Mobility Computer Adaptive Test (AM PAC CAT) score (month 6 minus baseline) and the [95% confidence interval] for patients assigned to each arm regardless of compliance are reported below. The AM PAC CAT is an item response theory-modeled scale that ranges from 0 to infinity. However, the score range of interest for the trial that corresponds to the ability to ambulate and transfer safely and independently (+/- gait aid) is 55 - 66 with higher scores corresponding to better mobility and the MID for improvement being 1.0. For the primary outcome group differences will be assessed over the 6 months of the trial using mixed-effects model repeated measures (MMRM) analysis which will include a random effect for patient, a fixed effect for measurement point (3 months or 6 months), and adjustment for age, gender, baseline value of the outcome variable, cancer type, cancer stage (IV versus other), and time.

SECONDARY OUTCOMES:
Pain as measured using the Brief Pain Inventory average and total pain interference subscales from baseline [6 months]. | From baseline to 6 months
  The change in the Brief Pain Inventory (BPI) average score and total interference score (Month 6 minus baseline) and the and the [95% confidence interval] for patients assigned to each arm regardless of compliance. The BPI average is a single numerical rating scale (NRS) anchored at 0 and 11. The total inference score is a composite of 6 NRS scales. Higher scores indicate more pain or a worse health state. For both measures the minimally important difference (MID) is population dependent and ranges between 0.5 and 2.0. For the secondary outcome group differences will be assessed over the 6 months of the trial using mixed-effects model repeated measures (MMRM) analysis which will include a random effect for patient, a fixed effect for measurement point (3 months or 6 months), and adjustment for age, gender, baseline value of the outcome variable, cancer type, cancer stage (IV versus other), and time.
Health Utility, as measured by the change in EuroQol 5-D (5Q-5D) scale score from baseline | From baseline to 6 months
  The change in health utility, as measured by the change in EuroQol 5-D (5Q-5D) score from baseline score (Month 6 minus baseline) and the and the [95% confidence interval] for patients assigned to each arm regardless of compliance. The EuroQol 5-D utility ranges from 0 to 1.0 with high values indicating better health states. The minimally important difference (MID) is population dependent and range between 0.5 and 1.0. For the secondary outcome group differences will be assessed over the 6 months of the trial using mixed-effects model repeated measures (MMRM) analysis which will include a random effect for patient, a fixed effect for measurement point (3 months or 6 months), and adjustment for age, gender, baseline value of the outcome variable, cancer type, cancer stage (IV versus other), and time.
Hospitalization frequency | From registration to 6 months
  The count of hospital admission lasting >24 hours. To assess the impact on number of hospitalizations we will use a negative binomial model, with an offset for number of days of follow-up.
Hospital length of stay | From registration to 6 months
  The count of days spent in the hospital for admissions lasting >24 hours. For patients who had at least one hospitalization, the impact of the interventions on the total number of days in hospital will be assessed using mixed effect Poisson analysis.
Discharge location from hospital | From registration to 6 months
  Binary variable describing whether patients were discharged to an inpatient facility (skilled nursing facility, inpatient rehabilitation facility, hospice or long term acute care facility) or home with/without services. Logistic models with random effects for patient will be used to analyze inter-group differences.
Planned admission | From registration to 6 months
  Binary variable describing whether an admission was planned for anti-cancer treatment or unplanned. Logistic models with random effects for patient will be used to analyze inter-group differences.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cheville, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Cheville AL, Moynihan T, Basford JR, Nyman JA, Tuma ML, Macken DA, Therneau T, Satelel D, Kroenke K. The rationale, design, and methods of a randomized, controlled trial to evaluate the effectiveness of collaborative telecare in preserving function among patients with late stage cancer and hematologic conditions. Contemp Clin Trials. 2018 Jan;64:254-264. doi: 10.1016/j.cct.2017.08.021. Epub 2017 Sep 5. PMID 28887068
- [Background] Cheville AL, Moynihan T, Herrin J, Loprinzi C, Kroenke K. Effect of Collaborative Telerehabilitation on Functional Impairment and Pain Among Patients With Advanced-Stage Cancer: A Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):644-652. doi: 10.1001/jamaoncol.2019.0011. PMID 30946436
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials